CLINICAL TRIAL: NCT03461770
Title: Continuous Positive Airway Pressure Decreased Lung Collapse During General Anesthesia Induction in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUS IV
Record Dates: First submitted 2018-02-14; First posted 2018-03-12 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-02

CONDITIONS: Atelectasis
Keywords: atelectasis; children; ultrasound
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients will receive anesthesia induction with Sevoflurane using a circular circuit without CPAP. Protective ventilation with 5 cmH20 of positive end-expiratory pressure (PEEP) will be initiated after induction. At the end of surgery, mechanical ventilation will stop allowing spontaneous ventilation. Patients will be extubated without CPAP. Lung ultrasound examinations will be performed at different times-points: before anesthesia induction, during surgery, at the end of surgery and before extubation, and after extubation.
- CPAP group (Experimental): Patients will receive anesthesia induction using 5 cmH20 of CPAP until the moment of intubation. After induction patients will receive the same protective ventilation than the control group. A lung recruitment maneuver will be applied if these patients present atelectasis during surgery. At the end of surgery, patients will be extubated under the modality of CPAP with 5 cmH20. Lung ultrasound examinations will be performed at different times-points: before anesthesia induction, during surgery, at the end of surgery and before extubation, and after extubation.
  Interventions: Other: CPAP

INTERVENTIONS:
Other: CPAP — Patients will receive general anesthesia induction with CPAP at 5 cmH20 via face mask with a circular system. CPAP will use before extubation.The air-test will perform during anesthesia with transitory decreases inspired fraction of oxygen to 0.21 over a 5 min period. Recruitment maneuver will be perform if the air test is positive, ( SpO2 is ≤ 96%)
  Arms: CPAP group

SUMMARY:
Anesthesia-induced atelectasis is a well-known entity observed in approximately 68-100% of pediatric patients undergoing general anesthesia. Infants and young children are more susceptible to this lung collapse due to their small functional residual capacity. Thus, intrapulmonary shunting caused by those atelectasis are more likely to occur during general anesthesia in infants and younger children than in adults. This problem predisposes children to hypoxemic episodes that can persist in the early postoperative period. Beyond the negative impact of atelectasis on gas exchange, mechanical ventilation induces a local inflammatory response in atelectatic lungs, even in healthy patients undergoing general anesthesia.

Therefore, the diagnosis, prevention and active treatment of anesthesia-induced atelectasis are mandatory, not only to avoid hypoxemic episodes and atelectasis-related post-operative pulmonary complications, but also to protect the lungs during mechanical ventilation. Nowadays, the diagnosis of anesthesia-induced atelectasis is easily and accurately accomplished by lung ultrasound (LUS). LUS is a simple and non-invasive tool useful to detect atelectasis in children, to assess lung aeration and for monitoring ventilator settings or strategies. Regarding to the prevention of atelectasis, it was demonstrated that the application of continuous positive airway pressure (CPAP) during the induction of general anesthesia decreases atelectasis formation in adult morbidly obese patients.

The investigators hypothesized that the use of CPAP during general anesthesia induction in pediatric patients can prevent or decrease atelectasis formation.

DETAILED DESCRIPTION:
Compare lung aeration between two different strategies of induction to general anesthesia: breathing throughout a facial mask without CPAP and breathing with 5 cmH20 of CPAP in pediatric patients scheduled for surgery under general anesthesia, using ultrasound imaging and a four-point-aeration score to assess the lung aeration.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by parents.
* Patients aged 6 months to 7 years old
* Scheduled for surgery under general anesthesia with tracheal intubation.
* American Society of Anesthesiologists classification: physical status I-II

Exclusion Criteria:

* Acute airway infection
* Cardiovascular or pulmonary disease
* Previous thoracic procedure

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Lung aeration during anesthesia | intraoperative
  Compare lung aeration between two different strategies of induction to general anesthesia: breathing throughout a facial mask without CPAP and breathing with 5 cmH20 of CPAP in pediatric patients scheduled for surgery under general anesthesia, using ultrasound imaging and a four-point-aeration score to assess the lung aeration (0 = normal lung, 1 = moderate aeration loss, 2 = severe aeration loss, 3 = complete aeration loss and consolidation).

SECONDARY OUTCOMES:
Peripheral arterial oxygenation by pulse oximetry | intraoperative
  Peripheral capillary oxygen saturation (SpO2) by pulse oximetry will be recorded during intra-operative anesthesia with the 'Air-Test'.
Lung aeration after surgery | immediately after surgery
  Lung aeration score immediately after surgery, using ultrasound imaging and a four-point-aeration score to assess the lung aeration (0 = normal lung, 1 = moderate aeration loss, 2 = severe aeration loss, 3 = complete aeration loss and consolidation).

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Acosta, MD, Principal Investigator — Hospital Privado de Comunidad
Locations (1):
- Cecilia M. Acosta, Mar del Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Acosta CM, Lopez Vargas MP, Oropel F, Valente L, Ricci L, Natal M, Suarez Sipmann F, Tusman G. Prevention of atelectasis by continuous positive airway pressure in anaesthetised children: A randomised controlled study. Eur J Anaesthesiol. 2021 Jan;38(1):41-48. doi: 10.1097/EJA.0000000000001351. PMID 33009190